CLINICAL TRIAL: NCT06906458
Title: Effect of Paresthesia During Interscalene Block Procedure on the Incidence of Postoperative Neurological Symptoms: A Prospective Observational Clinical Study
Brief Title: Impact of Paresthesia on Postoperative Neurological Symptoms
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Other Study IDs: Paresthesia
Record Dates: First submitted 2025-03-25; First posted 2025-04-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Interscalene Block; Postoperative Pain
Keywords: Interscalene block; Paresthesia; Postoperative neurological symptoms
MeSH Terms: conditions — Pain, Postoperative; Paresthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paresthesia: Patients experiencing paresthesia during the interscalene nerve block
  Interventions: Other: Paresthesia
- No paresthesia: Patients not experiencing paresthesia during the interscalene nerve block
  Interventions: Other: No paresthesia

INTERVENTIONS:
Other: Paresthesia — Patients experiencing paresthesia during the interscalene nerve block
  Groups: Paresthesia
Other: No paresthesia — Patients not experiencing paresthesia during the interscalene nerve block
  Groups: No paresthesia

SUMMARY:
In this study, the effect of paresthesia occurring during the interscalene block procedure on the incidence of postoperative neurological symptoms will be investigated. Paresthesia is defined as an abnormal sensation described as "tingling, pinprick, severe pain, or an electric feeling in the arm." The status of postoperative neurological symptoms in patients at the end of the block's effective duration will be assessed through phone interviews, evaluating symptoms such as arm numbness, tingling, abnormal sensations, pain, and weakness.

DETAILED DESCRIPTION:
Our study includes patients aged 18-65 years with American Society of Anesthesiologists (ASA) physical status I or II who undergo interscalene nerve block prior to arthroscopic shoulder surgery under general anesthesia. All patients will be fasting according to standard protocol. During the preoperative period, patients' age, comorbidities, gender, body mass index (BMI), ASA scores, and preoperative Quality of Recovery-15 (QoR-15) scores will be recorded.

In the operating room, possible complications related to the block (paresthesia, Horner's syndrome, dyspnea, hoarseness) will be monitored in the preoperative area. During the intraoperative period, data such as pulse, blood pressure, infusion fluids, intraoperative remifentanil requirements, anesthesia duration, and surgical time will be recorded.

In the postoperative period, postoperative pain status, block duration, postoperative nausea and vomiting, need for rescue analgesics and antiemetics, and QoR-15 scores on the first day will be assessed in the recovery room and ward. Additionally, postoperative neurological symptoms and QoR-15 scores will be followed via telephone on the 3rd, 7th, 10th, and 30th days after discharge.

For patients developing postoperative pain, pain intensity will be evaluated using an 11-point numeric rating scale, where 0 indicates no symptoms and 10 represents maximum severity.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I to II
* Age range of 18-65 years
* Patients planned for interscalene nerve block for analgesia prior to arthroscopic shoulder surgery in the beach chair position under general anesthesia

Exclusion Criteria:

* body mass index >35 kg/m²)
* history of drug use
* Patient's refusal to participate in the study
* Psychiatric disorders
* Central nervous system diseases
* Vestibular disorders
* Presence of diabetes, neuropathy, and paralysis
* Pregnancy
* Open shoulder surgery
* Allergy to local anesthetics
* Coagulopathy
* Severe thrombocytopenia
* Infection at the puncture site
* Pre-existing neuropathy in the limb to be operated on
* Use of opioid and antiemetic medications before surgery
* Use of dexamethasone
* Lung disease
* Low baseline oxygen saturation
* Patients who cannot cooperate in the postoperative period (e.g., mental retardation, delirium, language acquisition deficiency, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients aged 18-65 years with ASA physical status I or II who are planned to undergo interscalene nerve block for analgesia prior to arthroscopic shoulder surgery in the beach chair position under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Paresthesia incidence | Perioperative time
  Paresthesia is considered an abnormal sensation described as "tingling, pinprick, severe pain, or an electric feeling in the arm." When paresthesia occurs, the block procedure will be halted, and the needle will be redirected; local anesthetic will not be administered until the paresthesia resolves, and the occurrence of paresthesia will be recorded.

SECONDARY OUTCOMES:
Incidence of postoperative neurological symptoms | 30 days
  the status of postoperative neurological symptoms will be assessed via telephone by a physician different from the one who performed the block. During the evaluation, symptoms such as arm numbness, tingling, abnormal sensations, pain, and weakness will be considered. Those responding "yes" to any of these symptoms will be classified as patients experiencing postoperative neurological symptoms.
Postoperative pain | 36 hours
  In the postoperative period, patients will be assessed for pain using a 0-10 Numeric Rating Scale (NRS) at rest at 4, 6, 8, 12, 16, and 18 hours, and at both rest and during movement at 24 and 36 hours to record the highest pain scores. The NRS is a scale used for patients to express their pain levels, where 0 represents the absence of pain and 10 represents the most severe pain.
Duration of block effectiveness | 36 hours
  The time (in minutes) until the patient reports a significant increase in pain after the block
Postoperative nausea and vomiting | 36 hours
  Significant nausea, vomiting, and/or need for rescue antiemetics
Rescue analgesic requirement | 36 hours
  Number of additional analgesic applications
Rescue antiemetic requirement | 36 hours
  Number of additional antiemetic applications
intraoperative opioid requirement | intraoperative time
  To maintain the bispectral index (BIS) between 40-60, remifentanil will be initiated and titrated between 0.05-0.25 mcg/kg/min, taking into account a 20% increase in MAP (mean arterial pressure) compared to the initial value and a 15% increase in heart rate compared to the initial value.
Duration of stay in the recovery room | 2 hours
  The time from arrival in the recovery room until the discharge criteria are met
Quality of Recovery-15 (QoR-15) scores | 30 days
  The QoR-15 questionnaire consists of 15 questions rated on a scale of 0 to 10, with a total score assessed out of 150. Results are classified as follows: above 135 is considered "excellent," 122-135 is "good," 90-121 is "fair," and below 90 is "poor.
Horner's syndrome | Perioperative/Periprocedural
  Miosis and ptosis of the ipsilateral pupil during the perioperative period.
Dyspnea | Perioperative/Periprocedural
  Breathing difficulty as described by the patient during the perioperative period.
Hoarseness | Perioperative/Periprocedural
  Voice changes described by the patient during the perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No